CLINICAL TRIAL: NCT07254273
Title: Effects of Boccia Exercises on Upper Extremity Muscle Thickness and Grip Strength in Hemiparetic Individuals: A Randomized Controlled Trial
Brief Title: Boccia Exercises and Upper Limb Muscle Adaptations in Hemiparetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Emre Berk HAZAR, Research Assistant, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-15604681-100-234561
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hemiparesis After Stroke
Keywords: Stroke; ultrasound; upper extremity; hemiparatic; muscle thickness
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Interventional Study Model:
  Design: Randomized Controlled, Parallel Assignment, Pretest-Posttest Design Allocation: Randomized Intervention Model: Parallel Assignment Masking: Single (Outcomes Assessor) Primary Purpose: Treatment / Rehabilitation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boccia Exercise Group (Experimental): Participants in this group will receive conventional physical therapy combined with Boccia exercises three times per week for 8 weeks. Each session lasts approximately 45-60 minutes and includes warm-up, Boccia skill drills (target aiming, throwing control), and cool-down activities.
  Interventions: Other: Boccia exercise; Other: physiotherapy
- Control Group (Active Comparator): Participants in this group will receive only conventional physical therapy three times per week for 8 weeks. The program includes strengthening, range of motion, and task-specific functional exercises matched in duration and frequency to the experimental group.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: Boccia exercise — Boccia exercises differ significantly from other rehabilitation interventions for individuals with physical disabilities. Traditional physical therapy or exercise programs often involve repetitive, motivating movements that lack motivation and cannot be directly linked to individuals' daily activities. However, thanks to its game-based structure, Boccia offers a fun and functional exercise platform. This increases individuals' motivation to participate, facilitates continuity, and brings a more natural setting to the rehabilitation process. Furthermore, Boccia supports the active use of upper extremity muscles and the development of balance and coordination, while also encouraging social interaction and a sense of competition. Therefore, Boccia's game-based and accessible structure offers a more applicable and sustainable approach to developing motor skills and increasing functional independence in individuals with physical disabilities compared to other traditional interventions.
  Arms: Boccia Exercise Group
Other: physiotherapy — Conventional physical therapy (physiotherapy) is a proven rehabilitation approach aimed at improving upper extremity function, muscle strength, and range of motion in hemiparetic individuals who have had a stroke. The program includes strengthening exercises, joint mobilization, task-oriented functional activities, and motor relearning techniques. Sessions are individualized and tailored to the participant's clinical condition to increase independent participation in activities of daily living in hemiparetic individuals. Regular and structured practice helps prevent the development of muscle atrophy and contractures and maximize functional gains.

SUMMARY:
This study investigates whether adding Boccia exercises to conventional rehabilitation improves upper extremity muscle thickness and grip strength in individuals with hemiparesis following stroke. The research aims to determine if Boccia training can enhance muscle morphology and functional strength beyond standard physical therapy.

DETAILED DESCRIPTION:
Loss of upper extremity function after stroke significantly reduces independence in daily living. Changes in muscle morphology (muscle thickness, echogenicity, pennation, etc.) can affect strength, coordination, and functional performance. Boccia is a sport originally designed for individuals with special needs, encouraging hand-eye coordination, targeting, and force-controlled repetitions. Due to these characteristics, it has been suggested that boccia may positively impact both motor control and muscle tone; however, its effects on muscle morphology and grip strength in hemiparetic individuals have been limitedly studied. This study will investigate the contribution of boccia exercises to conventional physiotherapy on upper extremity muscle thickness and grip strength.

Primary objective: To evaluate whether boccia exercises provide significant improvements in upper extremity muscle thickness and grip strength after hemiparesis, in addition to conventional physical therapy.

Hypothesis: Participants who receive up to nine weeks of extended or eight weeks (8 weeks in the protocol) of boccia practice will show greater improvements in upper extremity muscle thickness and grip strength than those who receive conventional physical therapy alone.

This study is a parallel-group, random assignment controlled trial. The total sample included 22 stroke (hemiparetic) individuals; participants were randomly assigned to two groups: Boccia + physical therapy (Boc, n = 12) and physical therapy alone (Ctrl, n = 10). Assessments will be conducted at pre-intervention (baseline) and post-intervention (after 8 weeks). Assessors will be blinded to the measurements; complete blinding of operators and participants is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75
* Having had a stroke within the last 6-24 months and diagnosed with hemiparesis
* Mild to moderate motor function loss in the upper extremity (e.g., Fugl-Meyer Upper Extremity Score ≥ 20/66)
* Clinically stable individuals eligible to participate in sessions
* Be conscious, cognitively able to follow instructions, and consent
* Be physically fit enough to participate in exercise at least 3 days a week

Exclusion Criteria:

* Limited upper extremity movement due to severe spasticity, contracture, or joint deformity (Modified Ashworth Scale ≥ 3)
* Contraindication to exercise due to severe cardiovascular, pulmonary, or systemic disease
* Serious diseases other than neurological disorders (e.g., Parkinson's, MS, tumor)
* History of upper extremity surgery or trauma within the last 6 months
* Inability to exercise due to severe pain, infection, or skin lesions
* Inability to follow instructions due to psychiatric or cognitive impairment
* Concurrent participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
upper extremity muscle thickness | 8 weeks
  Muscle thickness of selected upper extremity muscles (e.g., biceps brachii, triceps brachii, deltoid) is measured using ultrasonography. Measurements are taken at standard anatomic locations with the participant in a relaxed, resting position. Thickness is recorded in millimeters (mm) and represents the distance between the superficial and deep aponeuroses of the muscle. Assessments are performed before (baseline) and after (8 weeks) the intervention by blinded assessors to assess changes in muscle morphology.

SECONDARY OUTCOMES:
Grip Strength | 8 weeks
  Maximum voluntary grip strength of the affected hand is measured using a hand dynamometer. Participants are seated with the elbow flexed at 90° and the forearm in neutral position. Three trials are performed, with brief rest periods between attempts, and the highest value (in kilograms, kg) is recorded. Assessments are conducted pre-intervention (baseline) and post-intervention (after 8 weeks) by blinded assessors to evaluate changes in upper extremity functional strength.

CONTACTS AND LOCATIONS:
Overall Officials: EMRE B HAZAR, Master Degree, Principal Investigator — Bayburt University
Locations (1):
- Bayburt Unıversity, Bayburt, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant privacy and comply with ethical and legal regulations.

REFERENCES:
- Available data/document: Individual Participant Data Set: The individual participant dat — https://docs.google.com/spreadsheets/d/1ZN1TbLb_kPid_fZNsQVWYNu02qO5s-mv/edit?usp=sharing&ouid=107542558214893941575&rtpof=true&sd=true — https://docs.google.com/spreadsheets/d/1ZN1TbLb_kPid_fZNsQVWYNu02qO5s-mv/edit?usp=sharing&ouid=107542558214893941575&rtpof=true&sd=true

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07254273/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT07254273/ICF_001.pdf